CLINICAL TRIAL: NCT03430479
Title: Phase Ib/II Study to Assess Efficacy, Safety & Immunological Biomarker of Anti PD-1 Antibody With Radiation Therapy in Patients With HER2-negative Metastatic Breast Cancer
Brief Title: Anti PD-1 Antibody With Radiation Therapy in Patients With HER2-negative Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kyoto Breast Cancer Research Network (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: kbcrnb002
Record Dates: First submitted 2018-02-06; First posted 2018-02-13 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental)
  Interventions: Drug: Cohort A
- Cohort B (Experimental)
  Interventions: Drug: Cohort A

INTERVENTIONS:
Drug: Cohort A — Radiation + Nivolumab + hormone therapy

SUMMARY:
The aim of this study is to evaluate the safety and efficacy of anti PD-1 antibody with radiation therapy in patients with HER2-negative metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

- Cohort A

1. Documentation of ER-positive and/or PR-positive tumor (>=1% positive stained cells) .
2. Patients must satisfy the following criteria for prior therapy:

   - Progressed during treatment or within 12 months of completion of adjuvant hormone therapy.

   or Progressed while prior hormone therapy for advanced/metastatic breast cancer. Two previous line of hormone therapy for advanced/metastatic disease is allowed.
3. Patients who have hormone therapy that can be expected for advanced /metastatic disease.

   Cohort B
4. Patients who have come to be non-responsive more than two line of chemotherapy
5. Prior chemotherapy with anthracycline and taxane agent

   Cohort A and B
6. Female patients who are histologically or cytologically confirmed to have breast cancer
7. Patients who have distant metastatic lesion as follow

   - More than one bone lesion for radiation therapy
8. Patients with cancer confirmed to be HER2-negative.（
9. Patients with a measurable lesion based on RECIST 1.1.
10. Patients aged >= 20 years at informed consent
11. Patients with ECOG PS of 0 to 1.
12. Patients without any severe disorder in the major organs.
13. Patients expected to survive for ≥ 90 days.
14. Patients of childbearing potential must be using an acceptable method of contraception to avoid pregnancy and must not be breastfeeding for 18 weeks after the last dose of investigational product
15. Patients who have provided written informed consent themselves.

Exclusion Criteria:

-

Exclusion Criteria:

1. Patients who have neuropathy (more than Grade 2)
2. Patients with any active autoimmune disease or a history of known autoimmune disease.
3. Patients who has a history of pneumonitis or interstitial lung disease.
4. Active, untreated central nervous system metastasis.
5. Patients with pericardial effusion, pleural effusion or ascites requiring treatment
6. Patients with uncontrolled diabetes mellitus
7. Patients with a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 28 days of the enrollment.
8. Patients who has received radiotherapy within 28 days of study registration, or radiotherapy for thorax within 56 days of the enrollment.
9. Pregnant or breast-feeding women.
10. Prior therapy with Nivolumab, anti CTLA-4 antibody therapies, any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
11. Patients considered ineligible for participation in this study by their attending physicians

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Phase Ib : dose-limiting toxicity rate | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Kyoto University Hospital, Kyoto, Japan

REFERENCES:
- [Derived] Takada M, Yoshimura M, Kotake T, Kawaguchi K, Uozumi R, Kataoka M, Kato H, Yoshibayashi H, Suwa H, Tsuji W, Yamashiro H, Suzuki E, Torii M, Yamada Y, Kataoka T, Ishiguro H, Morita S, Toi M. Phase Ib/II study of nivolumab combined with palliative radiation therapy for bone metastasis in patients with HER2-negative metastatic breast cancer. Sci Rep. 2022 Dec 27;12(1):22397. doi: 10.1038/s41598-022-27048-3. PMID 36575361